CLINICAL TRIAL: NCT06689605
Title: Ultrasound-guided Tru-cut Biopsy in Patients with Suspected Ovarian Cancer: Adequacy, Accuracy, Safety and Patient Assessment.
Acronym: TRUCUTOC
Status: Recruiting | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Other Study IDs: 202411 P05
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; tru-cut biopsy; expert ultrasonography
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A small amount of tissue from a tru-cut biopsy from ovarian cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective observational study is to evaluate the role of ultrasound-guided tru-cut biopsy (in the hands of an expert certified sonographer within a gynecological center)in patients with suspected ovarian cancer.

The main questions it aims to answer are:

Is the material from tru-cut biopsy adequate for histopathological and immunohistochemical examination? Is the material accurate in comparison with the final pathological specimen? What are the patient experience and complications after the procedure?

Participants who will undergo a standard tru-cut biopsy procedure will need to additionally answer the questionnaire.

DETAILED DESCRIPTION:
1. Current State of Knowledge

   Ovarian cancer remains the most lethal gynecologic malignancy, largely due to the lack of early detection and its presentation at a late stage1,2. In patients with ovarian cancer, the most important prognostic factor is the absence of macroscopic tumor at the end of surgery as well as the histological type3. For this purpose, adequate imaging before surgery, as well as histological knowledge of the tumor before the application of neoadjuvant chemotherapy is of great essence. Ultrasound-guided or CT-guided tru-cut biopsy in patients with advanced ovarian cancer has slowly become the preferred method of histological verification over the last decade in patients with suspected advanced ovarian cancer, with prof. Fischerová and her team being the pioneers in its use4,5.

   Our aim is to prospectively evaluate the role of ultrasound-guided tru-cut biopsy in the hands of an expert certified sonographer within a gynecological oncological center and with the material examined by a concrete expert in the gynecological oncological pathology field. The novelty in our approach so to say will lie in these three factors: prospective design, two expert sonographers, and one expert pathologist. This project will also be the first to include a patient experience survey after the procedure. Furthermore, with this project, we will be able to create a prospective database allowing for further work in the future.
2. Material Support for the Project

   The ultrasound examination will be performed on the GE Voluson E10 system located in the gynecological oncology center, tru-cut biopsy will be performed using a fast-gun automated biopsy system for sampling with 16-18 Gauge tru-cut needle and a G/16-30 cm core-cut biopsy needle. Histological examination will be performed in the state of art Fingerland department of pathology.
3. Project Objectives

   The goal of this project is to assess the adequacy of the material obtained from ultrasound-guided tru-cut biopsy for histopathological and immunohistochemical examination, compare for the accuracy of the histopathological diagnosis in samples with adequate material using the definitive surgical specimen as the reference standard while prospectively registering patient experience and complications after the procedure.
4. Methodology

All patients suspected of gynecological malignancies are regularly examined in the gynecological oncology tumor board. Patients with suspicion of advanced ovarian cancer will be indicated by the oncologist team member for expert ultrasound and tru-cut biopsy, these patients will be consecutively screened into the study after acquiring informed consent, patients who refuse consent will be monitored outside the study database. All patients will undergo coagulation tests before, including the appropriate management of anticoagulation treatment 6. The target population will be 30-40 patients over a period of two years.

Included patients will undergo expert ultrasound examination by two project members including both transabdominal and transvaginal examination using the International Ovarian Tumor Analysis (IOTA) and Morphological Uterus Sonographic Assessment (MUSA) terms. Before the tru-cut biopsy, a Doppler examination will be performed with the frequency set to define surrounding blood vessels. A 16-18 gauge tru-cut needle will be used. The transabdominal (freehand) or/and transvaginal (needle guide) approach to the biopsy will be performed by one project member using a 16-18 gauge tru-cut needle with the penetration depth set at 15-22mm. The biopsy will be repeated 2-3 times to acquire 2-3 samples for histopathological examination.

Following the procedure, patients will be observed for two hours in an outpatient setting for bleeding or early complications. Minor or major complications will be reported if they occur using the modified Dindo classification. A simple pain assessment survey will be filled in by the patient before dismissal. The biopsy material will be fixed in formalin and sent to the expert pathologist team member, results will be available within 3-5 working days. During the follow-up visit, another pain assessment survey will be filled to show the chronic effect after tru-cut biopsy. The patient will be examined again by the tumor board and after definitive surgery, the definitive material will be sent to the same expert pathologist who will be blinded to the initial diagnosis allowing for a blind reference standard.

All the data will be collected in three Excel databases and managed by three team members, one for histopathological information, one for ultrasound information, and one for safety and pain assessment. For statistics purposes, we will collect information on true positive, true negative, false positive, and false negative results. This will allow for the analysis of sensitivity, specificity, positive predictive value, and negative predictive value of the accuracy of ultrasound-guided tru-cut biopsy in patients with suspicion of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* suspected advanced ovarian cancer
* indication for tru-cut biopsy by multidisciplinary oncoboard

Exclusion Criteria:

* patient deny to undergo tru-cut biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected advanced ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adequacy of tru-cut biopsy in ovarian cancer | From the tru-cut biopsy to the histopathological result.
  Evaluation of the adequacy of the procedure in diagnosing ovarian cancer by histopathological and immunohistochemical examination.

SECONDARY OUTCOMES:
Accuracy of tru-cut biopsy in ovarian cancer | From the tru-cut biopsy to the definitive histopathological examination from the surgery.
  Evaluation of accuracy between tru-cut biopsy and definitive histology in ovarian cancer.

OTHER OUTCOMES:
Patient assesment | From the tru-cut biopsy to the first follow-up visit.
  To evaluate the patient experience with tru-cut biopsy and to record complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Undecided